CLINICAL TRIAL: NCT01859351
Title: A Phase I Open-label, Dose-escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of the PI3K Inhibitor WX-037, Given as a Single Agent and in Combination With the MEK Inhibitor WX-554, in Patients With Solid Tumors
Brief Title: Phase I Study of WX-037 Alone and in Combination With WX-554 in Solid Tumours
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated for business reasons
Sponsor: Heidelberg Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WX/90-001; 2012-004552-11 (EudraCT Number)
Record Dates: First submitted 2013-04-23; First posted 2013-05-21 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WX-037 (Experimental): PI3K inhibitor
  Interventions: Drug: WX-037
- WX-037 in combination with WX-554 (Experimental): PI3K inhibitor in combination with MEK inhibitor
  Interventions: Drug: WX-037; Drug: WX-554

INTERVENTIONS:
Drug: WX-037
Drug: WX-554
  Arms: WX-037 in combination with WX-554

SUMMARY:
The purpose of this study is to test the safety of escalating doses of the novel PI3K inhibitor WX-037 and to explore its effectiveness in combination with WX-554 which targets mitogen activated protein kinase (MEK1 and MEK2). Preclinical evidence indicates that these two novel compounds could provide targeted inhibition of both pathways to block tumour growth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced, metastatic and/or progressive solid tumors for whom there is no effective standard therapy available (for part 2 in addition patients for whom their PI3K pathway is deregulated)
* Evaluable or measurable disease
* Has normal organ function; is no greater than 2 on the ECOG performance scale
* Negative hCG test in women of childbearing potential

Exclusion Criteria:

* History of diabetes requiring daily medication or history of grade 3 or more fasting hyperglycemia
* Patients with major surgery, radiotherapy, or immunotherapy within 4 weeks of starting the study
* Clinical significant, unresolved toxicity from previous anti-cancer therapy
* Patients who previously received a MEK inhibitor (for combination part only)
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs
* Known medical history of retinal vein occlusion, intraocular pressure greater than 21 mm Hg or patient considered at risk of retinal vein thrombosis (combination part only)
* Known HIV positivity or active hepatitis B or C infection
* History of clinically significant cardiac condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose limiting toxicities | during cycle 1 (21days) of treatment with WX-037
Incidence of Dose Limiting toxicities | during cycle 1 (21 days) of treatment with WX-037 and WX-554

SECONDARY OUTCOMES:
Number of patients with adverse Events and serious adverse events | from cycle 1 day 1 until treatment discontinuation, an estimated average of 18 weeks
Assessment of PK variables, peak plasma concentration (Cmax), area under the curve (AUC) | two PK profiles in cycle 1
Determination of PD markers; changes from baseline in biomarkers of pathway inhibition | predose until treatment discontinuation, an estimated average of 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Udai Banerji, MD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Guy's and St Thomas' Foundation Trust, Guy's Hospital, London